CLINICAL TRIAL: NCT07318740
Title: The Effect of Mobile Application Supported Education and Counselling on Intention, Attitude, Behaviour and Self-Efficacy of Pregnant Women With Gestational Diabetes
Brief Title: Effectiveness of Mobile Application-Supported Education and Counseling in Pregnant Women With Gestational Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Gulhane Faculty of Nursing
Record Dates: First submitted 2025-08-26; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-08

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: Gestational Diabetes; Nursing; Mobile Application; Motivation; Self-Efficacy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Application-Based Education and Counseling (Experimental): Participants will receive a two-week structured education and counseling program via the SugarMoms mobile application for gestational diabetes management. The program, delivered by a certified diabetes nurse educator, covers topics including gestational diabetes management, blood glucose monitoring, insulin therapy, management of hypoglycemia and hyperglycemia, nutrition, physical activity, and pregnancy health recommendations. Each module includes audio support, a question-and-answer component, and daily motivational notifications (e.g., exercise, diet, hydration). Participants will record their daily blood glucose, dietary intake, and physical activity in the app. After completing the two-week program, participants will continue daily use of the app during the study. Follow-up assessments and questionnaires will also be administered through the app. Progress, logs, and module completion will be monitored via the administrator panel.
  Interventions: Behavioral: Mobile Application-Based Education and Counseling Program
- Standard Face-to-Face Gestational Diabetes Education (Active Comparator): Participants will receive a two-week standard face-to-face gestational diabetes education program provided by a certified diabetes nurse educator in accordance with the hospital protocol. The content will parallel the topics included in the intervention group's mobile application program. Blood glucose monitoring will be recorded using paper-based forms.
  Interventions: Behavioral: Standard Face-to-Face Gestational Diabetes Education

INTERVENTIONS:
Behavioral: Mobile Application-Based Education and Counseling Program — A two-week structured education and counseling program delivered via the SugarMoms mobile application for gestational diabetes management. Education is provided by a certified diabetes nurse educator and includes topics such as gestational diabetes management, blood glucose monitoring, insulin therapy, management of hypo/hyperglycemia, healthy nutrition, physical activity, and pregnancy health recommendations. Each module includes audio support, a question-and-answer component, and daily motivational notifications. Participants will log daily blood glucose, dietary intake, and physical activity in the app and continue app use throughout the study. Follow-up assessments and questionnaires are delivered through the app, and progress is monitored via the administrator panel.
  Arms: Mobile Application-Based Education and Counseling
Behavioral: Standard Face-to-Face Gestational Diabetes Education — A two-week standard face-to-face gestational diabetes education program provided by a certified diabetes nurse educator in accordance with hospital protocol. The program covers the same topics as the intervention group's app-based program. Blood glucose monitoring is recorded using paper-based forms.
  Arms: Standard Face-to-Face Gestational Diabetes Education

SUMMARY:
This randomized controlled trial aims to evaluate the impact of mobile application-supported education and counseling on the intention, attitude, behavior, and self-efficacy of pregnant women diagnosed with gestational diabetes. The study will be conducted at Ankara Bilkent City Hospital, with participants assigned to intervention and control groups. The intervention group will receive planned education and counseling via a mobile application, while the control group will receive standard hospital education. Data will be collected at predetermined intervals, and outcomes will be compared between the groups. The study seeks to determine the effectiveness of a mobile application-supported approach in the management of gestational diabetes.

DETAILED DESCRIPTION:
Gestational Diabetes Mellitus (GDM) is a carbohydrate intolerance disorder that develops during pregnancy or is first diagnosed during this period. If not properly managed, it can lead to serious complications for both the mother and the fetus. Current guidelines recommend healthy nutrition, regular physical activity, self-monitoring of blood glucose, and support from healthcare professionals for the management of GDM. In recent years, mobile health applications have emerged as valuable tools for providing pregnant women with rapid access to information, personalized counseling, and behavioural change support. However, studies evaluating the effects of mobile application-supported interventions in pregnant women with GDM who have initiated insulin therapy remain limited.

This randomized controlled trial aims to evaluate the effect of mobile application-supported education and counseling on the intention, attitude, behaviour, and self-efficacy levels of pregnant women with GDM who have initiated insulin therapy. The study will be conducted at the Internal Medicine Outpatient Clinic of the Obstetrics and Gynecology Hospital, Ankara Bilkent City Hospital. Pregnant women meeting the inclusion criteria will be randomly assigned to either the intervention or control group using a simple randomization method. A total of 94 participants (47 in the intervention group and 47 in the control group) will be included in the study.

In the intervention group, the developed mobile application will be installed on participants' smartphones, and a structured two-week education and counseling program will be implemented. The educational content will comprise seven modules: Essential Knowledge on Gestational Diabetes, Blood Glucose Monitoring in Pregnancy, Fundamental Information on Insulin Therapy in Pregnancy, Management of hypoglycemia and Hyperglycemia in Gestational Diabetes, Healthy Nutrition in Gestational Diabetes, Physical Activity and Exercise in Gestational Diabetes, and General Health Recommendations for a Healthy Life in Gestational Diabetes. Each educational module will be supported with audio recordings and followed by a question-and-answer session to enhance motivation. Daily motivational notifications (e.g., exercise reminders, healthy eating recommendations, water intake reminders) will be sent via the application, and participants' blood glucose records and module completion status will be monitored by the researcher through the administrator panel.

The control group will receive standard face-to-face diabetes education, in line with hospital protocols, for two weeks. This education will cover content comparable to that provided to the intervention group. Assessments will be conducted at three stages for both groups:

* Baseline assessment (before the start of education): Participant Identification Form, Gestational Diabetes Intention, Attitude, and Behaviour Scale, and Gestational Diabetes Self-Efficacy Scale.
* Second follow-up (three weeks after completion of the two-week education program): The same scales will be administered again.
* Third follow-up (two weeks after the second follow-up assessment): The Gestational Diabetes Intention, Attitude, and Behaviour Scale and the Gestational Diabetes Self-Efficacy Scale will be administered again. Additionally, the Mobile Health Applications Adoption Scale will be applied to the intervention group.

Throughout the study, all participants will be asked to regularly complete the Self-Monitoring of Blood Glucose (SMBG) log, whereas the intervention group will additionally record their blood glucose measurements via the mobile application. This study aims to generate robust evidence on the effectiveness of mobile health applications in managing GDM and to contribute to the wider adoption of digital health solutions during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women aged ≥18 years.

Minimum education level: primary school graduate.

Singleton pregnancy.

No prior diagnosis of gestational diabetes mellitus (GDM).

Newly diagnosed with GDM based on oral glucose tolerance test (OGTT) results.

Currently receiving insulin treatment as part of the clinical management plan.

Absence of comorbid conditions such as hypertension, preeclampsia, or other chronic diseases.

Ability to read and understand Turkish.

Ownership of a smartphone (iOS/Android) with internet access.

Willingness to participate and provide written informed consent.

Exclusion Criteria:

Development of pregnancy-related complications during the follow-up period.

Incomplete or missing data in the study forms.

Non-compliance with study protocol.

Withdrawal from the study at the participant's request.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Gestational Diabetes Intention, Attitude, and Behavior Scale (GDNTD-Ö) Scores | Baseline (before education), 3 weeks after completion of the 2-week education program (first follow-up), and 2 weeks after this first follow-up (second follow-up).
  This measure uses the validated Turkish adaptation of the Diabetes Intention, Attitude, and Behavior Scale. The instrument contains 14 items across 5 subdimensions. Total scores are transformed to a 0-100 scale, with higher scores indicating stronger intention, attitude, and behavior for self-management in gestational diabetes. There is no defined cut-off value. Measurement will be based on the self-administered GDNTD-Ö questionnaire.

SECONDARY OUTCOMES:
Change in Gestational Diabetes Self-Efficacy Scale (GESGD) Scores | Baseline (before education), 3 weeks after completion of the 2-week education program (first follow-up), and 2 weeks after this first follow-up (second follow-up).
  This measure consists of 23 items and 4 subdimensions (diet-weight management, complication prevention, adherence to nutrition education, and medical treatment practices). Higher scores indicate greater self-efficacy. There is no defined cut-off value. Measurement will be based on a self-administered questionnaire.

OTHER OUTCOMES:
Mobile Health Applications Adoption Scale Score (Intervention Group Only) | Second (final) follow-up, conducted 2 weeks after the first follow-up.
  This measure contains 31 items and 7 subdimensions, assessed on a 5-point Likert scale. Higher scores indicate greater adoption and acceptance of the mobile health application. This measure will be administered only to participants in the intervention group. Measurement will be based on a self-administered questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Gönül Kurt, Assoc. Prof. Dr., Principal Investigator — University of Health Sciences, Gülhane Faculty of Nursing, Department of Obstetrics and Gynecology Nursing
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared. Supporting documents such as the study protocol, statistical analysis plan, and informed consent form may also be provided.
Supporting Information: Study Protocol
Time Frame: 12 months after publication
Access Criteria: De-identified IPD will be available upon reasonable request to the Principal Investigator, conditional on signing a data sharing agreement.